CLINICAL TRIAL: NCT03879590
Title: Efficacy Of Doxophylline As A Sparing Treatment For Inhaled Corticosteroids In Mexican Children With Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Sandra Nora Gonzalez Diaz, Dra. med., Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DOXO
Record Dates: First submitted 2018-11-25; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Asthma Chronic; Asthma in Children
Keywords: doxophylline; asthma; steroid sparing
MeSH Terms: conditions — Asthma | interventions — doxofylline; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Budesonide and Doxophylline (Experimental): Budesonide at the same dose in which the subject is currently treated (GINA step 3 or 4) plus doxophylline at a dose of 18 mg / kg per day
  Interventions: Drug: Doxophylline; Drug: Budesonide
- Low budesonide and Doxophylline (Active Comparator): Reduced dose of inhaled budesonide (GINA step down) plus doxophylline to a dose of 18 mg / kg per day, maximum of 800 mg / day (Group B)
  Interventions: Drug: Doxophylline; Drug: Budesonide

INTERVENTIONS:
Drug: Doxophylline — Both groups will receive doxophylline one group will maintain the ICS dose and the other group will receive a reduced ICS dose (Maintaining the same GINA treatment step). After 4 weeks both groups will interchange treatment scheme.
  Other Names: There is no other intervention names
Drug: Budesonide — Both groups will receive doxophylline one group will maintain the ICS dose and the other group will receive a reduced ICS dose (Maintaining the same GINA treatment step). After 4 weeks both groups will interchange treatment scheme.
  Other Names: There is no other intervention names

SUMMARY:
This study evaluated the efficacy of doxophylline as a steroid sparing treatment in Mexican children with asthma treated with medium ir high doses of inhaled corticosteroids (ICS). It is a cross over study in which both groups of patients will receive doxophylline plus a lower steroid dose maintaining the same treatment step according to GINA guidelines, one group will maintain the same treatment dose while the other will start with doxophylline with the lower ICS dose, and by the middle of the study both groups will interchange treatment schemes.

DETAILED DESCRIPTION:
Inhaled corticosteroids (ICS) are first-line drugs for the treatment of persistent asthma. The effectiveness of existing ICS is excellent; however, a number of questions remain regarding its possible adverse effects, despite the fact that the use of the inhalation route has allowed the minimization of the systemic exposure to these drugs. Methylxanthines are widely used in the treatment of asthma. It is one of the few medications for asthma that can be administered orally. They are useful especially in patients who cannot adapt to inhaled medications. Methylxanthines are unique in exhibiting dual-function properties by inducing bronchodilation and having anti-inflammatory and immunomodulatory effects. Theophylline is the oldest methylxanthine and non-specifically inhibits phosphodiesterase, it is a little used drug because it has many adverse effects with lower therapeutic index. Doxophylline is a drug of the family of methylxanthines, with a similar efficacy compared to theophylline when applied in the treatment of various respiratory diseases, but with better tolerability profile. Doxophylline has been shown to be a bronchodilator and anti-inflammatory drug with a wider therapeutic window than other methylxanthines. Clinical studies have reported that doxophylline is more effective in improving lung function tests in adults and children, as well as in decreasing clinical symptoms, reducing the incidence of adverse effects and the need of emergency bronchodilators, with a better profile in terms of safety and it has been demonstrated that doxophylline potentially reduces the need for corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

1. Mexican patients between 6 and 16 years old.
2. Clinical diagnosis of asthma according to the current guidelines of the Global Asthma Initiative (GINA) 2018.
3. Patients with asthma treated with budesonide at medium or high doses during (GINA guidelines´ steps 3 or 4) at least two months before the first study visit. Budesonide medium dose: 200-400 mcg / day (6-11 years) and 400-800 mcg / day (> 12 years). Budesonide high dose: > 400 mcg / day (6-11 years) and > 800 mcg / day (> 12 years).

Exclusion Criteria:

1. Patients <6 or ≥16 years of age.
2. Patients with <16 kg of body weight.
3. Patients who have had an asthma exacerbation that required treatment with systemic corticosteroids (oral, intramuscular or intravenous) during the 2 months prior to the first study visit.
4. Patients who have presented an asthma exacerbation that required hospitalization during the 2 months prior to the first study visit.
5. Any other chronic lung disease that could impair lung function evaluation.
6. Cardiovascular, infectious, metabolic or neoplastic disease that could interfere with the evaluation of the patient.
7. Current use of drugs that interact with doxophylline: other xanthines, ephedrine or other sympathomimetics, erythromycin, troleandomycin, lincomycin, clindamycin, allopurinol, cimetidine, two months prior vaccination, propranolol, phenytoin or other anticonvulsants.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the values of the forced expiratory volume on the first second | 4 weeks
  Changes in the values of FEV1 (FEV1 in percent predicted) by comparing the baseline to subsequent evaluations.

SECONDARY OUTCOMES:
Use of rescue therapy | 4 weeks
  The use of rescue therapy defined as daily average of inhalations per day according to the data collected in the patient's diaries.
Clinical asthma control assessment | 4 weeks
  Differences in clinical asthma control assessment with a visual analogue scale (minimum score is 1, maximum score is 10,) comparing the baseline to follow-up evaluations.
Asthma exacerbations | 4 weeks
  Number of asthma exacerbations defined as acute episodes of progressively worsening shortness of breath, coughing, wheezing, and chest tightness or any combination thereof for at least 3 days, reported on the patient´s symptoms log.
Use of systemic corticosteroids | 4 weeks
  - The use of systemic corticosteroids for at least 3 days for the treatment of an asthma exacerbation according to the data collected in the patient's diaries.
Changes on the exhaled breath temperature | 4 weeks
  -Differences in values exhaled breath temperature measured in Celsius degrees with the X-halo device, comparing the baseline to follow-up evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Nora González-Díaz, PhD, Principal Investigator — Universidad Autónoma de Nuevo León

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lal D, Manocha S, Ray A, Vijayan VK, Kumar R. Comparative study of the efficacy and safety of theophylline and doxofylline in patients with bronchial asthma and chronic obstructive pulmonary disease. J Basic Clin Physiol Pharmacol. 2015 Sep;26(5):443-51. doi: 10.1515/jbcpp-2015-0006. PMID 25894641
- [Background] Margay SM, Farhat S, Kaur S, Teli HA. To study the efficacy and safety of doxophylline and theophylline in bronchial asthma. J Clin Diagn Res. 2015 Apr;9(4):FC05-8. doi: 10.7860/JCDR/2015/12438.5743. Epub 2015 Apr 1. PMID 26023566
- [Background] Rajanandh MG, Nageswari AD, Ilango K. Assessment of various second-line medications in addition to inhaled corticosteroid in asthma patients: a randomized controlled trial. Clin Exp Pharmacol Physiol. 2014 Jul;41(7):509-13. doi: 10.1111/1440-1681.12239. PMID 24738981
- [Result] Riffo-Vasquez Y, Venkatasamy R, Page CP. Steroid sparing effects of doxofylline. Pulm Pharmacol Ther. 2018 Feb;48:1-4. doi: 10.1016/j.pupt.2017.10.008. Epub 2017 Oct 16. PMID 29031617
- [Result] Rajanandh MG, Nageswari AD, Ilango K. Pulmonary function assessment in mild to moderate persistent asthma patients receiving montelukast, doxofylline, and tiotropium with budesonide: a randomized controlled study. Clin Ther. 2014 Apr 1;36(4):526-33. doi: 10.1016/j.clinthera.2014.02.006. Epub 2014 Mar 17. PMID 24650447

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03879590/Prot_SAP_000.pdf